CLINICAL TRIAL: NCT04512326
Title: RISK FACTORS FOR ANASTOMOTIC LEAKAGE FOLLOWING TOTAL OR SUBTOTAL COLECTOMY (RIALTCOT)
Acronym: RIALTCOT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Juan Ocaña Jiménez, Principal Investigator, Hospital Universitario Ramon y Cajal
Other Study IDs: 212/20
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Total Colectomy; Subtotal Colectomy
Keywords: Total colectomy; Subtotal colectomy; Ileorectal anastomosis; Ileosigmoid anastomosis; Anastomotic leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total or subtotal colectomy: Total or subtotal colectomy with ileorectal or ileosigmoid anastomosis
  Interventions: Procedure: Total or Subtotal colectomy

INTERVENTIONS:
Procedure: Total or Subtotal colectomy — Total or subtotal colectomy (emergent or elective) with primary anastomosis (ileorectal or ileosigmoid)

SUMMARY:
Higher anastomotic leakage (AL) rate is reported after ileosigmoid (ISA) or ileorectal anastomosis (IRA) in total or subtotal colectomy (TSC) compared to colonic or colorectal anastomosis. An AL reduction in these cases may improve short and long terms outcomes significantly. Current evidence remains insufficient to assess AL risk after TSC, based on single-center studies or small cases series. The investigators aim to analyse and identify potential risk factors to AL following TSC and ISA or IRA, both preoperative and intraoperative in order to prevent surgical complications.

The study is set up as a retrospective multicentre observational study. Inclusion criteria are patients (1) over 18 years old, (2) underwent restorative TSC with ISA or IRA anastomosis, (3) with/without loop ileostomy (4) between 2013-2019. Exclusion criteria are: (1) non-restorative TSC, (2) previous colorectal resection, (3) deferred anastomosis in trauma surgery and (4) other surgical resection in the same procedure.

AL will be defined as a defect of the integrity of the intestinal wall at the anastomotic site leading to a communication of the intra and extraluminal or a pelvic abscess adjacent to the anastomosis according to the definition set by de International Study Group of Rectal Cancer. AL requiring no active therapeutic intervention will be classified as Grade A. AL requiring active therapeutic intervention (antibiotics and percutaneous drainage) but manageable without relaparotomy will be classified as Grade B and AL requiring re-intervention were classified as Grade C.

Multivariable logistic regression model will be used in order to assess potential AL risk factors. p value <0,05 will be consider to indicate statistical significance.

Primary outcome is to assess potential risk factors to AL after restorative (ISA or IRA) TSC. Secondary outcomes are to identify risk factors to associated postoperative morbidity, mortality and re-admissions.

Data will be collected in each participating center enrolled in the study by the assigned principal investigator, confidentially and codified. Data will be sent to the study principal investigator. Database, patients code and email address will be provided at the study inclusion.

DETAILED DESCRIPTION:
Ileorectal (IRA) or ileosigmoid anastomosis (ISA) following Total or Subtotal Colectomy (TSC) are frequently performed in inflammatory bowel disease (IBD) (Crohn´s disease, ulcerative colitis and indeterminate colitis), familiar adenomatous polyposis or colonic polyposis syndromes and colorectal cancer (CRC). TSC is less frequently performed in refractory constipation and ischemic colitis.

Anastomotic leakage (AL) is a significant complication associate with increased mortality, reoperation and derivative morbidity and is also related to poor long term outcomes in oncological resections. Although, the formation of IRA or ISA is anatomically easy to performed, pelvic dissection is not mandatory, there is no tension at the anastomosis and a blood supply is theoretically ensured, higher AL risk is reported after IRA or ISA (6.5-21%) compared to colonic or colorectal anastomosis with lower AL rate, mainly under 15%. Regardless of the indication, similar AL rates are seen after TSC in IBD (4-12%), polyposis (20%) and colon cancer (6-21%). Reducing AL rates might improve short, long term and functional outcomes after IRA or ISA There is not a wide evidence about determinants for AL following colectomy with IRA or ISA.

The impact of the anastomosis (ISA or ISA) on AL is controversial with no findings any in the most recent studies. Great number of studies have been published about risk factors for AL after colectomy, but the majority are focused in colorectal cancer patients. IRA or ISA results after TSC are mixed with other anastomosis sites and the reported results are hardly clear and conclusive.

For this reason, The investigators aim to assess potential risk factors to AL in restorative TSC, including every surgical main reason.

ELIGIBILITY:
Inclusion Criteria:

* (1) over 18 years old
* (2) underwent restorative TSC with ISA or IRA anastomosis (emergent or elective)
* (3) with/without loop ileostomy
* (4) between 2013-2019

Exclusion Criteria:

* (1) non-restorative TSC
* (2) previous colorectal resection
* (3) deferred anastomosis in trauma surgery and
* (4) other surgical resection in the same procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent total or subtotal colectomy with primary anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage | 90 days postoperatively
  AL requiring no active therapeutic intervention will be classified as Grade A. AL requiring active therapeutic intervention (antibiotics and percutaneous drainage) but manageable without relaparotomy will be classified as Grade B and AL requiring re-intervention will be classified as Grade C

SECONDARY OUTCOMES:
Risk factors associated to postoperative morbidity | 90 days postoperatively
  Morbidity by Clavien-Dindo scale
Risk factors associated to mortality | 90 days postoperatively
  Mortality in postoperatively
Risk factors associated to re-admissions. | 90 days postoperatively
  Re-admissions after discharge within 90 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ocaña, MD, Principal Investigator — H.U Ramon y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elton C, Makin G, Hitos K, Cohen CR. Mortality, morbidity and functional outcome after ileorectal anastomosis. Br J Surg. 2003 Jan;90(1):59-65. doi: 10.1002/bjs.4005. PMID 12520576
- [Result] Moszkowicz D, Mariani A, Tresallet C, Menegaux F. Ischemic colitis: the ABCs of diagnosis and surgical management. J Visc Surg. 2013 Feb;150(1):19-28. doi: 10.1016/j.jviscsurg.2013.01.002. Epub 2013 Feb 20. PMID 23433833
- [Result] Washington C, Carmichael JC. Management of ischemic colitis. Clin Colon Rectal Surg. 2012 Dec;25(4):228-35. doi: 10.1055/s-0032-1329534. PMID 24294125
- [Result] Bakker IS, Grossmann I, Henneman D, Havenga K, Wiggers T. Risk factors for anastomotic leakage and leak-related mortality after colonic cancer surgery in a nationwide audit. Br J Surg. 2014 Mar;101(4):424-32; discussion 432. doi: 10.1002/bjs.9395. PMID 24536013
- [Result] Mirnezami A, Mirnezami R, Chandrakumaran K, Sasapu K, Sagar P, Finan P. Increased local recurrence and reduced survival from colorectal cancer following anastomotic leak: systematic review and meta-analysis. Ann Surg. 2011 May;253(5):890-9. doi: 10.1097/SLA.0b013e3182128929. PMID 21394013
- [Result] Law WL, Choi HK, Lee YM, Ho JW, Seto CL. Anastomotic leakage is associated with poor long-term outcome in patients after curative colorectal resection for malignancy. J Gastrointest Surg. 2007 Jan;11(1):8-15. doi: 10.1007/s11605-006-0049-z. PMID 17390180
- [Result] Lu ZR, Rajendran N, Lynch AC, Heriot AG, Warrier SK. Anastomotic Leaks After Restorative Resections for Rectal Cancer Compromise Cancer Outcomes and Survival. Dis Colon Rectum. 2016 Mar;59(3):236-44. doi: 10.1097/DCR.0000000000000554. PMID 26855399
- [Result] Duclos J, Lefevre JH, Lefrancois M, Lupinacci R, Shields C, Chafai N, Tiret E, Parc Y. Immediate outcome, long-term function and quality of life after extended colectomy with ileorectal or ileosigmoid anastomosis. Colorectal Dis. 2014 Aug;16(8):O288-96. doi: 10.1111/codi.12558. PMID 24428330
- [Result] 2015 European Society of Coloproctology Collaborating Group. Predictors for Anastomotic Leak, Postoperative Complications, and Mortality After Right Colectomy for Cancer: Results From an International Snapshot Audit. Dis Colon Rectum. 2020 May;63(5):606-618. doi: 10.1097/DCR.0000000000001590. PMID 32032201
- [Result] Platell C, Mackay J, Woods R. A multivariate analysis of risk factors associated with recurrence following surgery for Crohn's disease. Colorectal Dis. 2001 Mar;3(2):100-6. doi: 10.1046/j.1463-1318.2001.00213.x. PMID 12791002
- [Result] Nakamura T, Pikarsky AJ, Potenti FM, Lau CW, Weiss EG, Nogueras JJ, Wexner SD. Are complications of subtotal colectomy with ileorectal anastomosis related to the original disease? Am Surg. 2001 May;67(5):417-20. PMID 11379639
- [Result] Pastore RL, Wolff BG, Hodge D. Total abdominal colectomy and ileorectal anastomosis for inflammatory bowel disease. Dis Colon Rectum. 1997 Dec;40(12):1455-64. doi: 10.1007/BF02070712. PMID 9407985
- [Result] Loftus EV Jr, Delgado DJ, Friedman HS, Sandborn WJ. Colectomy and the incidence of postsurgical complications among ulcerative colitis patients with private health insurance in the United States. Am J Gastroenterol. 2008 Jul;103(7):1737-45. doi: 10.1111/j.1572-0241.2008.01867.x. Epub 2008 Jun 28. PMID 18564126
- [Result] Bjork J, Akerbrant H, Iselius L, Svenberg T, Oresland T, Pahlman L, Hultcrantz R. Outcome of primary and secondary ileal pouch-anal anastomosis and ileorectal anastomosis in patients with familial adenomatous polyposis. Dis Colon Rectum. 2001 Jul;44(7):984-92. doi: 10.1007/BF02235487. PMID 11496079
- [Result] Segelman J, Mattsson I, Jung B, Nilsson PJ, Palmer G, Buchli C. Risk factors for anastomotic leakage following ileosigmoid or ileorectal anastomosis. Colorectal Dis. 2018 Apr;20(4):304-311. doi: 10.1111/codi.13938. PMID 29059489